CLINICAL TRIAL: NCT03211143
Title: A Randomized, Open-label, Multiple-dose, and Crossover Study to Compare Pharmacokinetics, Pharmacodynamics and Safety of CKD-381 and D027 in Healthy Subjects
Brief Title: A Study to Compare PK, PD and Safety of CKD-381 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 173HPS16024
Record Dates: First submitted 2017-07-05; First posted 2017-07-07 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-06

CONDITIONS: GERD
Keywords: GERD; CKD-381; Nexium; Bioequivalence
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): TR group
  Period 1: Test drug(CKD-381), 1 tablet administered before the breakfast during 7 days
  Period 2: Reference drug(Nexium), 1 tablet administered before the breakfast during 7 days
  Interventions: Drug: CKD-381; Drug: Nexium
- B (Experimental): RT group
  Period 1: Reference drug(Nexium), 1 tablet administered before the breakfast during 7 days
  Period 2: Test drug(CKD-381), 1 tablet administered before the breakfast during 7 days
  Interventions: Drug: CKD-381; Drug: Nexium

INTERVENTIONS:
Drug: CKD-381 — Test drug: CKD-381
  Other Names: Esomeprazole 20mg+Sodum bicarbonate 800mg
Drug: Nexium — Reference drug: Nexium
  Other Names: Esomeprazole magnesium trihydrate 22.3mg

SUMMARY:
A Study to compare Pharmacokinetics, Pharmacodynamics and safety of CKD-381 and D027 in healty subjects

DETAILED DESCRIPTION:
A randomized, open-label, multiple-dose, and crossover study to compare pharmacokinetics, pharmacodynamics and safety of CKD-381 and D027 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Between 19 aged and 55 aged in healthy adult
2. Body weight more than 55kg in male, 50kg in female
3. Body Mass Index more than 18.5 and under 25(body mass index=kg/m2)
4. If female, must include more than one among the items

   * The menopause(there is no natural menses for at least 2 years)
   * Surgical Infertility(hysterectomy or bilateral oophorectomy, tubal ligation or other methods of infertility condition
5. If men has sexual life with women of childbearing age, Necessarily he agrees that use condoms and do not sperm donation until two months during clinical trials and after the final dosage of investigational products
6. Those who fully understand about this clinical trials after enough hearing, and then decided to join the clinical trials by themselves and to comply with the precautions written consent.

Exclusion Criteria:

1. Have clinically significant disease that hepatobiliary system(severe hepatic impairment, etc), kidney(severe renal impairment, etc), nervous system, immune system, respiratory system, endocrine system, hemato-oncology disease, cardiovascular system(heart failure, etc) or mental illness, or a history of mental disease.
2. Have a gastrointestinal disease history that can effect drug absorption(Crohn's disease, ulcers, etc.) or surgery(except simple appendectomy or hernia surgery)
3. Hypersensitivity reaction or clinically significant hypersensitivity reaction in the history of Esomeprazole, additives or benzimidazole family
4. Have a history of fructose intolerance, glucose-galactose malabsorbtion or sucrase isomaltase deficiency
5. Defined by the following laboratory parameters

   * Na>1.5 upper limit of normal range
   * AST, ALT>1.25 upper limit of normal range
   * Total bilirubin>1.5 upper limit of normal range
   * CPK>1.5 upper limit of normal range
   * eGFR(using by MDRD method)<60mL/min/1.73m2
   * Positive for HBV, HCV and HIV by serology test
   * Positive by urine drug abuse test.
   * Sitting SBP > 140mmHg or < 90mmHg, sitting DBP > 90mmHg or < 60mmHg, after 5 minutes break.
6. Have a history of drug abuse
7. Subject takes ethical drug or herbal medicine within 14 days, OTC within 7 days before the beginning of study treatment but investigator determine that the taking drug affect this study or could affect the safety of subjects.
8. Subject who takes inhibitor and inducers of drug metabolizing enzyme(Barbiturates etc.) within 30 days.
9. smoker(except the one who have stopped smoking more than 90days before beginning of study treatment)
10. A heavy caffeine consumer(caffeine>5 cups/day), alcohol consumer(alcohol>210g/week),
11. Taking foods containing grapefruit within 7 days before the beginning of study treatment(ex. Drinking containing grapefruit of 1L per a day or more within 7 days before the beginning of study treatment)
12. Subject who treated with any investigational drugs within 90 days before the beginning of study treatment
13. Previously donate whole blood within 60 days or component blood within 30 days.
14. Pregnant or lactating women.
15. An impossible one who participants in clinical trial by investigator's decision including laboratory test result or another reason

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics(Area under the plasma drug concentration-time curve within a dosing interval(AUCτ)) | 0h~12 h
  Evaluating PK of Esomeprazole after Multiple dose
Pharmacodynamics(Percent decrease from baseline in integrated gastric acidity for 24-hour interval after 7th dose) | Baseline versus Multiple dose during 7days
  Evaluating PD for ambulatory 24hr pH monitor

CONTACTS AND LOCATIONS:
Overall Officials: Choon Ok Kim, MD, Principal Investigator — Clinical Trials center, Yonsei Univ. Health system
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim D, Park MS, Yoo BW, Hong T, Park SJ, Kim CO. The safety, pharmacodynamics, and pharmacokinetics of immediate-release formulation containing esomeprazole 20 mg/sodium bicarbonate 800 mg in healthy adult male. Drug Des Devel Ther. 2019 Sep 3;13:3151-3159. doi: 10.2147/DDDT.S212491. eCollection 2019. PMID 31564831